CLINICAL TRIAL: NCT05329493
Title: A Novel Cooling Device for Pain Management During Fingerstick Blood Draw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dieter Manstein, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000271
Record Dates: First submitted 2022-03-29; First posted 2022-04-15 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Blood
Keywords: Blood Draw; Fingerstick Blood Draw

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cooling digit device application (Experimental): Device: Cooling digit device. The cooling finger device will be applied in the subjects on their right hand. Subjects will serve as their own control.
  Interventions: Device: Cooling digit device application

INTERVENTIONS:
Device: Cooling digit device application — Cooling digit device will be applied on subject's right hand ( fifth finger).
  Other Names: cooling finger device

SUMMARY:
In this study, the investigators seek to evaluate a novel tissue-cooling device for pain management during needle sticks and /or blood draw on the fingertips.

DETAILED DESCRIPTION:
Patient compliance with laboratory testing is one of the most underrecognized challenges in developing a treatment plan for acute and chronically ill patients. The ability to offer alternatives to standard venipuncture blood draws would greatly increase a laboratory's ability to provide testing to patients and health care providers.The fingerstick blood draw has been used as an alternative.

Aiming a less painful, potentially easier alternative we devised a novel that can be applied distally on the digit prior to the blood collection procedure and may provide analgesia through a liquid coolant that is run through tubes in the device to safely cool tissue to achieve numbing. We hypothesize that this device will safely and effectively reduce the pain associated with the fingertip pricks and increase the amount of capillary blood collected.

Multiple punctures with a large lancet were a frequent cause of discomfort among patients.With this new device the discomfort will be reduced by its application followed by the numbness of the finger.

The investigators plan to have 12 patients to complete the study. Subjects must be equal to greater than 18 years old and younger than 60 years older and may be any gender or Fitzpatrick skin type.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.

  * Male or Female subjects, ≥ 18 and ≤ 60 years of age at the time of enrollment.
  * All Fitzpatrick Skin Types are eligible
  * General good health confirmed by medical history and skin examination of the area to be treated
  * Subjects fifth finger is 17-23mm in diameter at the distal phalanges.

Exclusion Criteria:

* • Subject has had a surgical procedure(s) in the intended area of treatment in the last 6 months.

  * Sensitivity to the cold or history of cold-induced diseases including Raynaud's disease and cryoglobulinemia
  * Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
  * Suffering from significant skin conditions in treatment areas or inflammatory skin condition, including but not limited to open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Principal Investigator's discretion) or during the treatment course.
  * History of keloid scarring, abnormal wound healing and /or prone to bruising.
  * History of epidermal or dermal disorders (Particularly if involving collagen or micro vascularity) including collagen vascular disease or vasculitis disorders
  * Subject is unable or unwilling to comply with the study requirements.
  * Subject is currently enrolled or has been enrolled within the prior 3 months in a clinical study of any other unapproved investigational drug or device.
  * Any other condition that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Manstein, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Clinical Unit for Research Trials & Outcomes in Skin, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Jankowski CA, Casapao AM, Siller S, Isache C, Cani KV, Claudio AM, Brown M, Milstid B, Feldhammer M. Preanalytical Challenges During Capillary Fingerstick Sampling Preclude Its Widespread Use in Adult Hospitalized Patients. Am J Clin Pathol. 2021 Feb 11;155(3):412-417. doi: 10.1093/ajcp/aqaa138. PMID 33009571
- [Background] Kertes DA, Kamin HS, Liu J, Bhatt SS, Kelly M. Putting a finger on the problem: Finger stick blood draw and immunization at the well-child exam elicit a cortisol response to stress among one-year-old children. Psychoneuroendocrinology. 2018 Jul;93:103-106. doi: 10.1016/j.psyneuen.2018.04.021. Epub 2018 Apr 22. PMID 29705575
- [Background] Iwasawa H, Nishimura T, Nemoto S, Aikawa N, Watanabe K. Correlation of the Blood Test Results Obtained between Assays Using Microliter-scale Fingertip Blood Samples Collected with a Novel Blood Collection Device and Conventional Venous Blood Assays: a Secondary Publication in English. Keio J Med. 2018 Jun 25;67(2):26-34. doi: 10.2302/kjm.2017-0009-OA. Epub 2017 Nov 21. PMID 29162770
- [Background] Sugimoto S, Tateishi A, Osawa S. [Development of the fingertip blood dilution method for blood cell counting]. Rinsho Byori. 2014 Mar;62(3):235-40. Japanese. PMID 24800498

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: fingers
Groups:
- Cooling Digit Device Application: The cooling finger device will be applied to all study participants on their hand (fifth or third finger). The hand picked will be randomized and opposite to that of the control hand. Subjects will serve as their own control.
- Control: All study participants will have their fifth or third finger pricked. Subjects will serve as their own control.
Period: Overall Study
Arm/Group | Cooling Digit Device Application | Control
Started | 6; 6 fingers | 6; 6 fingers
Completed | 6; 6 fingers | 6; 6 fingers
Not Completed | 0; 0 fingers | 0; 0 fingers

BASELINE CHARACTERISTICS:
Arm/Group | Cooling Digit Device Application
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Wong-Baker FACES Pain Rating Scale
Description: This scale will be used to record subject pain from the overall pain from the procedure for the treatment and control finger. There are 6 faces ranging from 0 no hurt to 10 hurts the worst.
Time Frame: day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: fingers
Arm/Group | Cooling Digit Device Application | Control
Number analyzed (Participants) | 6 | 6
Number analyzed (fingers) | 6 | 6
score on a scale | 1.2 (0.8) | 2.4 (0.5)

2. Secondary Outcome: Blood Absorption Via Whatman 903 Filter Paper (Surface Area)
Description: After the finger has been pricked, the finger will subsequently be held over a single-use Whatman 903 filter paper. Approximately every ten seconds after the prick, the filter paper will be gently applied to the blood drop to absorb the blood. This will be repeated on new locations of the filter paper until blood flow stops. At least one Whatman 903 filter paper will be used per finger prick. The Whatman 903 filter paper will be imaged.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: cm^2
Units Other Than Participants: fingers
Arm/Group | Cooling Digit Device Application | Control
Number analyzed (Participants) | 6 | 6
Number analyzed (fingers) | 6 | 6
cm^2 | 1.4 (0.8) | 1.1 (0.7)

3. Secondary Outcome: Blood Absorption Via Whatman 903 Filter Paper (Drops of Blood)
Description: as for outcome 2
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: number of drops
Units Other Than Participants: fingers
Arm/Group | Cooling Digit Device Application | Control
Number analyzed (Participants) | 6 | 6
Number analyzed (fingers) | 6 | 6
number of drops | 11.4 (2.5) | 12.4 (8.4)

ADVERSE EVENTS:
Time Frame: 31 days
Description: Minimal-risk study with healthy participants. Evaluations were ongoing throughout the study to detect adverse events and changes in existing medical conditions.
Arm/Group | Cooling Digit Device Application | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT05329493/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT05329493/ICF_001.pdf